CLINICAL TRIAL: NCT07333027
Title: Effects of Loneliness in the Treatment of Depression
Brief Title: Lonely in Depression
Status: Recruiting | Type: Observational
Sponsor: Friedrich-Alexander-Universität Erlangen-Nürnberg (Other)
Collaborators: Bezirkskliniken Mittelfranken, Clinic for Psychiatry, Addiction, Psychotherapie and Psychosomatic Medicine, Am Europakanal, Germany (Unknown)
Responsible Party: Principal Investigator, Franziska Sonnauer, Dr. med. Franziska Sonnauer, Principal Investigator, Friedrich-Alexander-Universität Erlangen-Nürnberg
Other Study IDs: 25-435-B
Record Dates: First submitted 2025-12-02; First posted 2026-01-12 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Depression Disorder; Loneliness
Keywords: loneliness; depression; prospective; biosampling; clinical
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — Blood samples: EDTA and Serum collection --> blood, plasma, serum, cells (PBMCs, Leukocyten) Salvia samples: Salivette® Cortisol Stool samples: stool collection tubes with stabilizer --> microbiome analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this prospective study is to better understand the link between loneliness and depression in the inpatient psychiatric treatment of depression. It aims to answer:

Do lonely and not lonely persons benefit the same way from inpatient depression treatment? Is loneliness a clinical relevant factor in inpatient treatment of depression? What are the underlying biopsychosocial mechanisms?

Participants will be asked to do some

* self-report questionnaires
* clinical interview
* biosampling (blood, saliva, stool) at three main measurement timepoints (1. begin of inpatient treatment, 2. day of discharge, 3. three months after discharge).

DETAILED DESCRIPTION:
Loneliness and depression are widespread and severely debilitating health conditions. Notably, loneliness and depression are closely intertwined, with individuals suffering from depression being particularly vulnerable to loneliness. However, little is known regarding the clinical significance of loneliness in the treatment of depression and the biopsychosocial mechanisms underlying this association.

To examine the clinical relevance of the interplay between loneliness and depression, a prospective, noninterventional longitudinal design will be adopted. The study will be performed at the University Hospital and the community hospital in Erlangen, Germany. Every patient admitted to the hospital with depressive symptoms is eligible for screening according to the inclusion and exclusion criteria. Three main measurement points (T0, T1, and T2) and brief interim measurements conducted at two-week intervals (t0.1 to t0.X and t1.1-t1.6) will be utilized. After screening and clinical interviews, participants will complete the baseline measurements (T0). Thereafter, each participant will adhere to an individual period corresponding to the duration of that specific patient's inpatient stay at the clinic until the second measurement is obtained (T1). Follow-up will occur three months after T1.

Given that the effect sizes of the interaction between loneliness and depression in a clinical population are currently unknown, the sample size for this study was determined based on considerations of practicability and the population generalizability of the obtained results, as well as statistical plausibility.

To ensure the external validity of the results, it is important that both severely lonely depressive patients and less lonely depressive patients, as well as different disease trajectories and patient characteristics (e.g., age, sex, and number of comorbidities), can be identified. A sample size of approximately 200 participants is expected to ensure sufficient heterogeneity. This sample size is practically feasible due to the fact that, even when considering an inclusion rate of 50% and a dropout rate of 30% for the primary diagnosis of depression at the University Hospital and the community hospital in Erlangen, the recruitment potential clearly exceeds the target number of cases within an estimated period of two years.

Without the knowledge of which measured level of loneliness at baseline represents a strong level of loneliness and which measured level represents a weak level of loneliness in a depressed patient population, a median split of loneliness at baseline will be performed to calculate the statistical significance of the interaction between loneliness and depression in the inpatient and follow-up course (T0, T1, and T2). To detect a significant interaction effect of a mixed analysis of variance (ANOVA), when considering an α error of 0.05, a power of 0.9 (1-β error probability) and a correlation value among repeated measures of 0.5 for the groups defined as highly lonely and slightly lonely groups, the number of cases was calculated by using G*Power Version 3.1.9.7. Assuming a small effect size (f= 0.10), the desired sample size would be determined at n= 214 individuals; moreover, assuming a medium effect size (f= 0.25), the sample size would be n= 36 individuals. This indicates that there is statistical plausibility for detecting interaction effects between loneliness and depression with the target number of cases.

Eligibility screening and clinical diagnostic screening, along with interviews, are conducted by study physicians. Depression is assessed during a clinical interview (MADRS) by the patient's treatment team, which also determines when the patient will be discharged from the hospital. All of the self-report assessments are collected by the patients themselves by using the REDCap online survey application. Biosampling will be exclusively performed among participants recruited at the University Hospital to ensure methodologically consistent and rapid processing. Routine clinical data are primarily extracted from clinical documentation systems and consolidated prior to analysis (similar to other data sources).

Given that the study design does not permit definitive causal conclusions to be determined regarding the direction of effects, the findings are expected to provide valuable insights and relevant implications. In particular, the following insights can be obtained: (1) a report on whether more or less lonely patients receive equal benefits from inpatient multimodal depression treatment; (2) insights into changes in loneliness during and after depression treatment; (3) important findings regarding the shared and nonshared biopsychosocial mechanisms underlying loneliness and depression; and (4) the effects of loneliness and depression with respect to secondary outcomes, including quality of life and suicidality.

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis of depression according to ICD-10 (F32 or F33), as diagnosed by a physician or clinical psychologist in conjunction with the M.I.N.I. Mini-International Neuropsychiatric Interview diagnostic tools
* inpatient elective or emergency admission to one of the two psychiatric clinics; - age over 18 years
* sufficient understanding of spoken and written German
* informed voluntary consent

Exclusion Criteria:

* a current lack of capacity to provide consent (e.g., pronounced psychotic symptoms, stuporous depressive syndrome, and thought constriction to suicidality)
* previous participation in the study
* pregnancy or breastfeeding
* inpatient stay of less than 7 days, even if the patients initially met the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who are admitted for inpatient treatment at one of the two psychiatric clinics in Erlangen (university hospital, community hospital), Germany, either electively or as an emergency case, due to depressive symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-02-05 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Depression | Baseline/T0 (recruitment, normally day 1 of inpatient stay and maximum of day 4), T1 (end of inpatient stay, normally 7 days up to 50 weeks), Follow-Up/T2 (three months after clinical discharge); measured T0 to T1 and T0 to T2 and T1 to T2
  Montgomery-Åsberg Depression Rating Scale (MADRS) (10 Items, each item rated 0-6 points, minimum 0 points, maximum 60 points, higher scores indicate greater severity of depressive symptoms)
Loneliness | Baseline/T0 (recruitment, normally day 1 of inpatient stay and maximum of day 4), T1 (end of inpatient stay, normally 7 days up to 50 weeks), Follow-Up/T2 (three months after clinical discharge); measured T0 to T1 and T0 to T2 and T1 to T2
  3 Item UCLA Loneliness Scale (3-Item UCLA) (3 items, each item rated 1-3 points, minimum 3 points, maximum 9 points, higher scores indicate greater loneliness)
Depression | Baseline/T0 (recruitment, normally day 1 of inpatient stay and maximum of day 4), T1 (end of inpatient stay, normally 7 days up to 50 weeks), Follow-Up/T2 (three months after clinical discharge); measured T0 to T1 and T0 to T2 and T1 to T2
  Patient Health Questionnaire, 9-Item Depression Scale (PHQ-9) (9 Items, each item rated 0-4 points, minimum 0 points, maximum 27 points, higher scores indicate greater severity of depression)
Loneliness | Baseline/T0 (recruitment, normally day 1 of inpatient stay and maximum of day 4), T1 (end of inpatient stay, normally 7 days up to 50 weeks), Follow-Up/T2 (three months after clinical discharge); measured T0 to T1 and T0 to T2 and T1 to T2
  6-Item short scales for Loneliness, De Jong Gierveld Loneliness Scale (6-Item DJGLS) (6 Items, each item rated 1-3 points, before the total score is calculated, the items are dichotomized, thus resulting in a sum score ranging from 0 to 6, wherein scores of 0-1 indicate no loneliness, 2-4 indicate moderate loneliness, and 5-6 indicate severe loneliness)

SECONDARY OUTCOMES:
Social Support | Baseline/T0 (recruitment, normally day 1 of inpatient stay and maximum of day 4), T1 (end of inpatient stay, normally 7 up to 50 weeks), Follow-Up/T2 (three months after clinical discharge); measured T0 to T1 and T0 to T2 and T1 to T2
  Fragebogen zur Sozialen Unterstützung (F-SoZ-U 14) (14 Item shortend form, each item rated 0-4 points, minimum 0 points, maximum 56 points, higher total scores indicating higher levels of perceived social support)
Inpatient treatment duration | Baseline/T0 (recruitment, normally day 1 of inpatient stay and maximum of day 4) to T1 (end of inpatient stay, normally 7 up to 50 weeks).
  in days
Quality of life in self-report | Baseline/T0 (recruitment, normally day 1 of inpatient stay and maximum of day 4), T1 (end of inpatient stay, normally 7 days up to 50 weeks), Follow-Up/T2 (three months after clinical discharge); measured T0 to T1 and T0 to T2 and T1 to T2
  World Health Organization-Five Well-Being Index (WHO-5) (5 Items, each item rated 0-5 points, minimum 0 points, maximum 25 points, the total score (0-25) is transformed to a scale ranging from 0 to 100, with scores ≤50 indicating diminished well-being and higher scores representing higher well-beeing)
Social Network measure (newly designed for this study) | Baseline/T0 (recruitment, normally day 1 of inpatient stay and maximum of day 4), T1 (end of inpatient stay, normally 7 days up to 50 weeks), Follow-Up/T2 (three months after clinical discharge); measured T0 to T1 and T0 to T2 and T1 to T2
  As there is no culture and language adapted version of a social network indice available an adapted and German-translated version is used to capture participants' social interaction partners during the prior two weeks. The questionnaire was newly developed, with item content informed by existing validated scales (Cohen Social Network Index (SNI), Lubben Social Network Scale (LSNS), Berkman - Social Network/Integration).
  Via the use of a yes/no response format, participants indicated whether they had personal or telephone contact with each of the following: (1) spouse or partner, (2) own children, (3) parents or parent-like figures, (4) other relatives (e.g., siblings, uncles, or aunts), (5) friends, (6) neighbors, (7) colleagues, (8) people known through voluntary activities, (9) in-laws (parents, sons, or daughters-in-law), and (10) members of their social group (e.g., community, congregation, sports, or music clubs).
  Higher total scores indicate greater social connectedness.
General health status | Baseline/T0 (recruitment, normally day 1 of inpatient stay and maximum of day 4), T1 (end of inpatient stay, normally 7 days up to 50 weeks), Follow-Up/T2 (three months after clinical discharge); measured T0 to T1 and T0 to T2 and T1 to T2
  Short Form 12 Health Survey (SF-12) (12 Items, Items rated 0-1, 1-3 and 1-5 and 1-6 scores represent eight dimensions of physical and mental well-beeing with two composite scores, items are recodet, z-transformed and normed, higher values indicate better health)
Social Anxiety | Baseline/T0 (recruitment, normally day 1 of inpatient stay and maximum of day 4), T1 (end of inpatient stay, normally 7 days up to 50 weeks), Follow-Up/T2 (three months after clinical discharge); measured T0 to T1 and T0 to T2 and T1 to T2
  Social Phobia Inventory (SPIN) (17 Items, each item rated 0-4 points, minimum 0 points, maximum 68 points, higher scores indicate greater severity of social anxiety, three subscales are available (fear 6 items, avoidance 7 items, physiological distress 4 items))
Somatic Symptom Burden | Baseline/T0 (recruitment, normally day 1 of inpatient stay and maximum of day 4), T1 (end of inpatient stay, normally 7 days up to 50 weeks), Follow-Up/T2 (three months after clinical discharge); measured T0 to T1 and T0 to T2 and T1 to T2
  13-Item Somatic Symptom Severity Scale of the Patient Health Questionnaire (PHQ-13) (13 Items, each item rated 0-2 points, minimum 0 points, maximum 34 points, higher values indicating more somatic symptoms)

OTHER OUTCOMES:
Blood markers (metabolic, LDL) | Baseline/T0 (recruitment, normally day 1 of inpatient stay and maximum of day 4), T1 (end of inpatient stay, normally 7 days up to 50 weeks), Follow-Up/T2 (three months after clinical discharge); measured T0 to T1 and T0 to T2 and T1 to T2
  LDL cholesterin [mg/dl or mmol/l], higher values (> 100 mg/dl or > 2.6 mmol/l) represent unfavorable metabolic risk
Blood markers (metabolic, HDL) | Baseline/T0 (recruitment, normally day 1 of inpatient stay and maximum of day 4), T1 (end of inpatient stay, normally 7 days up to 50 weeks), Follow-Up/T2 (three months after clinical discharge); measured T0 to T1 and T0 to T2 and T1 to T2
  HDL cholesterin [mg/dl or mmol/l), < 40 mg/dl men and < 50 mg/dl women represents unfavorable metabolic risk, ≥ 40 mg/dl men ≥ 50 mg/dl women acceptable, ≥ 60 mg/dl protective
Blood markers (metabolic, HbA1c) | Baseline/T0 (recruitment, normally day 1 of inpatient stay and maximum of day 4), T1 (end of inpatient stay, normally 7 days up to 50 weeks), Follow-Up/T2 (three months after clinical discharge); measured T0 to T1 and T0 to T2 and T1 to T2
  HbA1c [%], higher values (> 5.7%) represent unfavorable metabolic risk
Blood markers (Sphingolipid metabolism) | Baseline/T0 (recruitment, normally day 1 of inpatient stay and maximum of day 4), T1 (end of inpatient stay, normally 7 days up to 50 weeks), Follow-Up/T2 (three months after clinical discharge); measured T0 to T1 and T0 to T2 and T1 to T2
  Sphingolipid metabolism enzyme activity of secretory acid sphingomyelinase (S-ASM) [nmol/mL/h/µL], higher leveles represent more inflammation/apoptosis enzyme activity of neutral acid sphingomyelinase (N-ASM) [nmol/mL/h/µL], higher levels represent cellular stress/apotosis Ceramide [nmol/L], higher levels represent more inflammation/apoptosis
Blood markers (neutrotrophic factor, BDNF) | Baseline/T0 (recruitment, normally day 1 of inpatient stay and maximum of day 4), T1 (end of inpatient stay, normally 7 days up to 50 weeks), Follow-Up/T2 (three months after clinical discharge); measured T0 to T1 and T0 to T2 and T1 to T2
  brain-derived neurotrophic factor [ng/mL], higher levels represent more neuroplasticity
Blood markers (hormonal) | Baseline/T0 (recruitment, normally day 1 of inpatient stay and maximum of day 4), T1 (end of inpatient stay, normally 7 days up to 50 weeks), Follow-Up/T2 (three months after clinical discharge); measured T0 to T1 and T0 to T2 and T1 to T2
  Cortisol [µg/dL or nmol/L] and timepoint of blood test higher levels represent more stress response
Blood markers (immunological markers) | Baseline/T0 (recruitment, normally day 1 of inpatient stay and maximum of day 4), T1 (end of inpatient stay, normally 7 days up to 50 weeks), Follow-Up/T2 (three months after clinical discharge); measured T0 to T1 and T0 to T2 and T1 to T2
  C-reactive protein (CRP) [mg/L], higher levels show systemic inflammation
Saliva marker (cortisol) | Baseline/T0 (recruitment, normally day 1 of inpatient stay and maximum of day 4), T1 (end of inpatient stay, normally 7 days up to 50 weeks), Follow-Up/T2 (three months after clinical discharge); measured T0 to T1 and T0 to T2 and T1 to T2
  saliva cortisol (awakening and before bedtime), higher levels represent more stress response
Saliva marker (α-amylase) | Baseline/T0 (recruitment, normally day 1 of inpatient stay and maximum of day 4), T1 (end of inpatient stay, normally 7 days up to 50 weeks), Follow-Up/T2 (three months after clinical discharge); measured T0 to T1 and T0 to T2 and T1 to T2
  saliva α-amylase activity [U/ml] (awakening and before bedtime), higher levels represent more stress response
Stool markers | Baseline/T0 (recruitment, normally day 1 of inpatient stay and maximum of day 4), T1 (end of inpatient stay, normally 7 days up to 50 weeks), Follow-Up/T2 (three months after clinical discharge); measured T0 to T1 and T0 to T2 and T1 to T2
  alpha-diversity
Suicidality (clinician rated) | Baseline/T0 (recruitment, normally day 1 of inpatient stay and maximum of day 4), T1 (end of inpatient stay, normally 7 days up to 50 weeks), Follow-Up/T2 (three months after clinical discharge); measured T0 to T1 and T0 to T2 and T1 to T2
  measures in clinical interview (Montgomery-Åsberg Depression Rating Scale (MADRS)) (Item No. 10 out of 10 items, rated 0-6, higher values represent more suicidality)
Suicidality (self-report) | Baseline/T0 (recruitment, normally day 1 of inpatient stay and maximum of day 4), T1 (end of inpatient stay, normally 7 days up to 50 weeks), Follow-Up/T2 (three months after clinical discharge); measured T0 to T1 and T0 to T2 and T1 to T2
  9-Item Patient Health Questionnaire (PHQ-9) (Item No. 9 out of 9, rated 0-3 with higher scores indicating more suicidality)
Response (depression) | Baseline/T0 (recruitment, normally day 1 of inpatient stay and maximum of day 4) to T1 (end of inpatient stay, normally 7 days up to 50 weeks).
  ≥ 50% reduction in Montgomery-Åsberg Depression Rating Scale (MADRS) score from T0 to T1 (10 Items, each item rated 0-6 points, minimum 0 points, maximum 60 points, higher scores indicate greater severity of depressive symptoms)
Relapse (depression) | T1 (end of inpatient stay/discharge from clinic) to Follow-Up/T2 (three months after clinical discharge).
  ≥ 10 points more from T1 to T2 in Montgomery-Åsberg Depression Rating Scale (MADRS) score or ≥ 22 points at T2 (10 Items, each item rated 0-6 points, minimum 0 points, maximum 60 points, higher scores indicate greater severity of depressive symptoms)
Antidepressant medication | Baseline/T0 (recruitment, normally day 1 of inpatient stay and maximum of day 4), T1 (end of inpatient stay, normally 7 days up to 50 weeks), Follow-Up/T2 (three months after clinical discharge); measured T0 to T1 and T0 to T2 and T1 to T2
  consideration of these classes of antidepressant drugs if these are given in a dosage that is effective as an antidepressant (e.g. for Mirtazapin not 7.5 mg, starting from 15 mg): SSRI/SNRI/NaSSA(Mirtazapin)/NDRI (Buproprion)/TZA/MAO-I/SARI (Trazodon)Agomelatin/other with classes of augmentation strategy: Lithium/antipsychotics/second antidepressant/other augmentation strategy sorted as: antidepressant monotherapy/antidepressant augmented therapy/other and change in therapy stategy (1. no; 2. yes drug substance (2.1) added/ (2.2) changed/ (2.3) removed; 3. yes dosage of antidepressant changed (3.1) increased/(3.2) decreased; 4. augmentation strategy changed)
trait vs. state loneliness | Baseline/T0 (recruitment, normally day 1 of inpatient stay and maximum of day 4), T1 (end of inpatient stay, normally 7 days up to 50 weeks), Follow-Up/T2 (three months after clinical discharge); measured T0 to T1 and T0 to T2 and T1 to T2
  Given the absence of an established measure capable of differentiating between enduring (trait) and situational (state) loneliness, this aspect is captured by using a newly developed single item: 'In looking back upon my life, I would say that I have felt …'. Participants respond to this item on a four-point scale (1= mostly lonely throughout my life, 2= lonely from time to time, 3= only lonely at present, and 4= never lonely). Responses of 1 are intended to represent trait loneliness; options 2 and 3 represent state loneliness; and option 4 indicates no loneliness.
number of therapies participated | Baseline/T0 (recruitment, normally day 1 of inpatient stay and maximum of day 4) to T1 (end of inpatient stay, normally 7 days up to 50 weeks).
  frequency per week of psychotherapy, group interventions and other

CONTACTS AND LOCATIONS:
Overall Officials: Franziska Sonnauer, Dr. med., M.Sc., Principal Investigator — Department of Psychiatry and Psychotherapy, Friedrich-Alexander Universität Erlangen-Nürnberg
Locations (2):
- Germany (2):
  - Friedrich-Alexander-Universität Erlangen-Nürnberg, Erlangen, Bavaria
  - Bezirkskliniken Mittelfranken, Clinic for Psychiatry, Addiction, Psychotherapie and Psychosomatic Medicine, Erlangen, Bavaria

IPD SHARING:
Plan to Share IPD: Undecided
IPD used in the results publication No final desicion has been made as several partners are involved and feasibility and regulatory requirements are still under review.